CLINICAL TRIAL: NCT01013636
Title: Epidemiology and Clinical Presentation of Human Anaplasmosis in Eastern France
Brief Title: Human Anaplasmosis in Eastern France
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER/ Directeur de la recherche clinique et des innovations, University Hospital, Strasbourg, France
Other Study IDs: 3960
Record Dates: First submitted 2009-11-10; First posted 2009-11-16 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Anaplasmosis; Tick-borne Disease; Ehrlichia
MeSH Terms: conditions — Anaplasmosis; Tick-Borne Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anaplasma
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — * Anaplasma diagnosis test : serology and PCR
  * If presence of Anaplasma infection, proposition of treatment with doxycylin 200 mg once-a-day during 10 days

SUMMARY:
Anaplasmosis is a tick-borne transmitted infection. Its clinical expression include fever, cytopenia and hepatitis.This infection was initially described in United States. In Europe, its epidemiology is not well known. Some isolated cases have been diagnosed in several country, were the tick Ixodes ricinus is known to transmitted another infection :the Lyme borreliosis.The purpose of our study is to look systematically for Anaplasmosis, in patient living in Eastern France, and presenting with compatible clinical symptoms using a new diagnosis tool : PCR in blood samples. So we will have new data about epidemiology in our country and the clinical symptoms that are associated with Anaplasmosis.

ELIGIBILITY:
Inclusion Criteria:

* patient with at least one of following symptoms : fever or muscular pain or articular pain or respiratory signs or neurological signs or meningitis or erythema occurring during the three weeks after a tick bite-
* Or
* patient with fever with at least one of following criteria : thrombocytopenia, leucopenia, hepatitis, without any other cause that can explain these abnormalities.
* Or
* patient with tick-borne encephalitis, or primary stage Lyme borreliosis

Exclusion Criteria:

* children less that 10 years
* pregnancy
* patients with an other diagnosis that can explain clinical symptoms or biological abnormalities
* antibiotherapy with cyclins during the days before inclusion

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Anaplasma phagocytophilia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Risk factor, clinical and biological markers of infection for patients with Anaplasma antibody seroconversion | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: YVES HANSMANN, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales Hôpitaux Universitaires de Strasbourg
Locations (12):
- France (12):
  - Service des Maladies Infectieuses et Tropicales - CHU de Besançon, Besançon
  - Centre Hospitalier de Colmar, Colmar
  - Département d'Infectiologie CHU de Dijon, Dijon
  - Centre Hospitalier de Guebwiller, Guebwiller
  - Centre Hospitalier de Haguenau, Haguenau
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Service des Maladies Infectieuses et Tropicales - CHU de Nancy, Nancy
  - Service de Médecine Interne et Maladies Infectieuses - CHU de Reims, Reims
  - Centre Hospitalier de Saverne, Saverne
  - Centre Hospitalier de Sélestat, Sélestat
  - Service des Maladies Infectieuses et Tropicales Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre hospitalier de Wissembourg, Wissembourg